CLINICAL TRIAL: NCT05357937
Title: The Impact of a Structured Physiotherapy Program on Pulmonary Function and Walking Capacity in Obese and Non-obese People Undergoing Cardiac Surgery
Brief Title: Structured Physiotherapy Program in Obese and Non-obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Dr. Mohammad Abu Shaphe, Associate Professor, University of Jazan
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ref No: 05/JUREC/14PT.2020
Record Dates: First submitted 2022-04-05; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Obesity
Keywords: Coronary artery bypass grafting; Obesity; Rehabilitation; Spirometry; Six Minute walk Test
MeSH Terms: conditions — Coronary Artery Disease; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese group (Active Comparator): Received standard physiotherapy program
  Interventions: Behavioral: standard physiotherapy program
- Non-Obese group (Active Comparator): Received standard physiotherapy program
  Interventions: Behavioral: standard physiotherapy program

INTERVENTIONS:
Behavioral: standard physiotherapy program — A qualified physical therapist administered a structured physiotherapy program from day 1 to day 7 in both groups

SUMMARY:
A routine physiotherapy program has been shown to be effective in the prevention and treatment of cardiopulmonary diseases. It also significantly increases functional capacity following coronary artery bypass grafting. However, the effect of a structured physiotherapy program in obese and non-obese patients has not been well explored. As such, the objective of this study is to determine the effect of a standardized physiotherapy program on pulmonary function and walking capacity in obese and non-obese patients undergoing coronary artery bypass grafting. A prospective study was conducted on 50 obese and non-obese individuals who were schedule for coronary artery bypass grafting. Their body mass index was used to separate them into two groups. Both groups followed a structured physiotherapy program from day 1 to day 7 post cardiac surgery. Both groups underwent spirometry and a six-minute walk test at baseline (preoperatively) and after day 4 and day 7 postoperatively. The effect of physiotherapy program on pulmonary function and 6-MWT was assessed using an independent t-test. To estimate the percentage increase or decrease of pulmonary function and distance during 6-MWT for obese and non-obese groups, the percent difference between baseline and posttest data was calculated and compared using an independent t-test. When the normality test failed, the Mann Whitney U test and analysis of variance on rank were used. Chi-square test was used for gender distribution. The results were considered statistically significant if p ≤ 0.05.

DETAILED DESCRIPTION:
METHODS Study participants and data collection The Research Ethics Committee of Jazan University, Saudi Arabia gave its approval to this study (Ref No: 05/JUREC/14PT.2020). Prior to participation, each participant signed an informed consent form. All experiments were carried out in line with the Helsinki Declaration. A prospective study was conducted on 50 consecutive individuals (26 obese, 24 non-obese). People aged 70 years or older, or who had any orthopedic or neurological difficulties were excluded from the trial. People were informed about the trial and consented in writing. Following enrollment, participants were placed into two groups according to their BMI. Participants in Group A were obese, defined as having a BMI of > 30 to < 35 kg/m2. Participants in Group B were non-obese, defined as having a BMI of > 25 to < 29.9 kg/m2.

Subjective ratings and spirometry data were taken at baseline. All spirometry tests were performed in the sitting position using the Vitalograph 2120 in accordance with established guidelines. At least three times, the readings were taken, and the best result was used. A posttest spirometry was performed on day 4 and 7 postoperatively. A six-minute walk (6-MWT) test was conducted at baseline and on day 7 postoperatively. Patients were advised to walk back and forth on the walking path at their own pace for 6-MWT. They were given six minutes to cover as much ground as possible. When 4 and 2 minutes remained in the test, prompts were offered. We utilized the following standardized prompt: "You're down to the final two (or four) minutes. You are doing an excellent job. You may accelerate or decelerate at any time, maintain the same pace, or take a break if necessary. Simply attempt to travel as much distance as possible in the remaining time. You are doing an excellent job." After six minutes, the participant's total distance traveled was recorded, along with a Borg dyspnea scale rating. A qualified physical therapist administered a structured physiotherapy program from day 1 to day 7 in both groups.

Statistical analysis The descriptive variables are expressed as mean ± standard deviation. The effect of physiotherapy program on pulmonary function and 6-MWT was assessed using an independent t-test. To estimate the percentage increase or decrease of pulmonary function and distance during 6-MWT for obese and non-obese groups, the percent difference between baseline and posttest data was calculated and compared using an independent t-test. When the normality test failed, the Mann Whitney U test and analysis of variance on rank were used. Chi-square test was used for gender distribution. The results were considered statistically significant if p ≤ 0.05. Statistical analyses were performed using the Statistical Package for Social Sciences (SPSS, Windows version-17.0, SPSS Chicago. IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Both obese and non-obese patient awaiting Coronary artery bypass graft

Exclusion Criteria:

* People aged 70 years or older, or who had any orthopedic or neurological difficulties were excluded from the trial.

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Mean changes in pulmonary function | day 7
  Pulmonary functions were measured using the spirometry tests in the Vitalograph 2120 in accordance with established guidelines. At least three times, the readings were taken, and the best result was used. A posttest spirometry was performed on day 4 and 7 postoperatively.
Mean changes in distance walked during six-minute walk test | day 7
  A six-minute walk (6-MWT) test was conducted at baseline and on day 7 postoperatively . Patients were advised to walk back and forth on the walking path at their own pace for 6-MWT. They were given six minutes to cover as much ground as possible. When 4 and 2 minutes remained in the test, prompts were offered. We utilized the following standardized prompt: "You're down to the final two (or four) minutes. You are doing an excellent job. You may accelerate or decelerate at any time, maintain the same pace, or take a break if necessary. Simply attempt to travel as much distance as possible in the remaining time. You are doing an excellent job." After six minutes, the participant's total distance traveled was recorded, along with a Borg dyspnea scale rating.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor, Principal Investigator — University of Jazan
Locations (1):
- Jazan University, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No